CLINICAL TRIAL: NCT07034521
Title: The Feasibility and Therapeutic Effect of Hybrid End-effector Robot-assisted Gait Training With an Active-assisted Module in Chronic Stroke Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202504096DSE
Record Dates: First submitted 2025-06-11; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Rehabilitation; Robotic Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- passive mode (Active Comparator)
  Interventions: Device: HIWIN MRG-P110
- active-assistive mode (Active Comparator)
  Interventions: Device: HIWIN MRG-P110

INTERVENTIONS:
Device: HIWIN MRG-P110 — HIWIN MRG-P110 is a robotics for lower limbs rehabilitation

SUMMARY:
Walking rehabilitation after stroke is most effective during the first three months of recovery, but even in the chronic phase-beyond six months post-stroke-a significant number of patients still show potential for gait improvement. Robot-assisted rehabilitation is becoming increasingly common in clinical settings, with various design modes available. However, the effectiveness of new products in improving gait or motor function still requires further investigation.

This study aims to evaluate the usability and therapeutic effects of a new end-effector exoskeleton robot system, HIWIN MRG-P110, for gait training in chronic stroke patients. The system uses foot pedal mechanisms to drive hip and knee movements for lower-limb training. Unlike its predecessor, this device allows adjustment of the active assistance ratio, encouraging users to engage in voluntary movement. It is designed for gait training in stroke patients and others with neurological impairments, but the usability and efficacy of this new training model remain to be verified.

This clinical trial is a randomized, single-blind, prospective study enrolling 60 stroke patients who are 6 months to 3 years post-onset and have a Functional Ambulation Category (FAC) level of 0 to 3. The study will explore how patients with varying degrees of motor weakness learn to adapt to the "active-assistive mode" in terms of speed and perception. Participants will be randomly assigned to either the active-assistive mode group or the fully passive mode group. Both groups will receive 15 treatment sessions over 5 weeks.

The study will compare the two groups in terms of:

1. Improvements in gait and balance immediately post-treatment and at 3-month follow-up
2. Changes in brain activity, as measured by functional near-infrared spectroscopy (fNIRS)

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years old.
* First-ever stroke, confirmed by brain CT or MRI, with onset between 6 months and 3 years prior to enrollment.
* Walking ability classified as Functional Ambulation Category (FAC) level 0 (non-ambulatory) to level 3 (able to walk short distances indoors or outdoors only).
* Prior to the current stroke, the participant was an independent community ambulator without mobility impairments.

Exclusion Criteria:

* Presence of lower limb joint contractures, deformities, or severe spasticity (Modified Ashworth Scale score of 4).
* Lower limb musculoskeletal conditions causing wounds, pain, inability to bear weight, or significant leg length discrepancy (>2 cm after orthotic correction).
* Known osteoporosis (T-score < -2.5) or history of osteoporotic fractures in the thoracolumbar spine or hip joints.
* Inability to use the exoskeleton device due to body size, including:

Body weight > 135 kg; Height < 145 cm or > 190 cm Thigh length < 38 cm or > 48 cm; Calf length < 48 cm or > 52 cm

* Cognitive or communication impairments that prevent understanding of study instructions or completion of questionnaires.
* Acute infections or unstable vital signs.
* Significant orthostatic hypotension or inability to maintain upright posture for more than 30 minutes.
* Use of indwelling urinary catheter, nasogastric tube, or tracheostomy.
* Pregnant women.
* Terminal illness with life expectancy less than six months.
* Inability to attend 15 rehabilitation sessions and follow-up assessment at 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
10 meter walk test | baseline, right after last session of intervension (within 1 week), 3 months after intervension

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No